



# **Ministry of Health**

Assessing SARS-CoV-2 Seroprevalence during Routine Antenatal Care Visits in Zambia

#### **Protocol Version 1.1**

## 13 June 2021

# **Principle and Co-Investigators**

| Affiliation | Name | Role |
|------------------------|-----------------------------|--------------|
| Zambia National Public | Muzala Kapina, MBChB (PI) | Protocol |
| Health Institute | Nyambe Sinyange, MBChB, MSc | development, |

| | John Simwanza, MBChB | implementation, |
|---|---|---|
| | Otridah Kapona, MSc | monitoring, data |
| | , | management and |
| | | analysis, report |
| | | writing |
| Ministry of Health | Lloyd Mulenga, MBChB, PhD, MMed (PI) | Protocol |
| | Sombo Fwoloshi, MBChB, MMed | development, |
| | Aaron Shibemba, MBChB, MMed | implementation, |
| | Kennedy Malama, MBChB, MPH | monitoring, data |
| | Powell Choonga, MSc | management and |
| | Angel Mwiche, MBChB, MMED | analysis, report |
| | Maureen Chisembele, MBChB, MMED | writing |
| | Consity Mwale, MBChB, MMED | |
| | Gideon Mwale, MBChB, MPH | |
| Centre for Infectious | Izukanji Sikazwe, MBChB, MPH (PI) | Protocol |
| Disease Research in | (CITI expiration: 9 Feb 2022) | development, |
| Zambia | Mwanza Wa Mwanza, MD | implementation, |
| | Carolyn Bolton, MBChB, MSc | monitoring, data |
| | Theodora Savory, MD | management and |
| | | analysis, report |
| | | writing |
| Centers for Disease | Jonas Hines, MD | Protocol |
| Control and Prevention | (CITI expiration: 2 January 2022) | development, |
| | Elizabeth Heilmann, MPH | implementation, |
| | (CITI expiration: 25 June 2023) | monitoring, data |
| | Adam Wolkon, MPH | management and |
| | (CITI expiration: 26 December 2021) | analysis, report |
| | Sam Yingst, DVM, PhD | writing |
| | (CITI expiration: 31 October 2022) | |
| | Warren Malambo, MPH | |
| | (CITI expiration: 11 February 2022) | |
| | Julie Gutman, MD MSc | |
| | (CITI expiration: 25 June 2022) | |
| | Laura Steinhardt, PhD, MPH | |
| | (CITI expiration: 19 January 2022) | |

**CDC's role:** CDC will not engage in data collection or have access to identifiable data; rather, CDC will provide technical leadership on protocol development, data collection procedures, data analysis, interpretation of results, and their dissemination. All data will be owned by the Zambia Ministry of Health.

**Funding source:** Buffer component COVID-19 response Cooperative Agreement number: NU2GGH002251, Provincial Ownership to Uplift Delivery of HIV/TB Services in Zambia (PROUD-Z) through technical Assistance

**Conflict of interest:** The primary investigators and co-investigators have no personal, financial, or other relationships that might pose a conflict of interest (or the appearance of a conflict) in their role in this activity. The contents in this protocol are those of the authors and do not necessarily represent the official position of the Centers for Disease Control and Prevention.

#### **Differences from CDC umbrella protocol**

This protocol was adapted from a generic protocol approved by CDC entitled, "Assessing COVID-19 seroprevalence from routine antenatal care visits," approved on 12/17/2020 (eClearance ID: 0900f3eb81c55548). No major methodological changes were made. Minor differences made in response to local feedback include:

- Prevalence estimates at district level rather than health facility level
- Twenty women each will be recruited from 40 health facilities among 4 districts each month compared to 30 women from 30 health facilities
- First visit ANC routine lab tests (HIV, syphilis, Hepatitis B, and/or malaria) will be recorded on the questionnaire
- Per guidance from the CDC-Atlanta team, several questions on potential exposure were removed from the questionnaire and COVID-19 vaccination history was added (compared to the generic protocol questionnaire)

# **Table of Contents**

| Α | Acronyms | .6 |
|---|---|---|
| 1.0 | Introduction | . 7 |
| 1 | .1 General information on research topic | .7 |
| 1 | 2 Overview of research and research gaps | .8 |
| 1 | 3 Overall purpose of the research | .8 |
| 2.0 | Statement of the Problem | .9 |
| 3.0 | Rationale/ Justification | .9 |
| 4.0 | Literature Review | .9 |
| 5.0 | Research questions | 10 |
| 6.0 | Research Aims and Objectives | 10 |
| 6 | 5.1 Research Aim | 10 |
| 6 | 3.2 Primary Objectives | 10 |
| 6 | 3.3 Secondary Objectives | 11 |
| 7.0 | Methodology | 11 |
| 7 | '.1 Study Design | 11 |
| 7 | '.2 Study Site and Population | 11 |
| 7 | '.3 Selection of Participants, Sampling and Sample Size | 13 |
| 7 | '.4 Implementation of Procedures | 15 |
| 7 | .5 Quality control and Assurance activities (supervisory, data and logistics monitoring) | 18 |
| 7 | '.6 Study staff roles and responsibilities | 19 |
| 7 | 7.7 Data collection and management | 20 |
| 7 | '.8 Data analysis | 21 |
| 7 | '.9 Data Ownership | 21 |
| 7 | '.10 Sponsor monitoring | 21 |
| 7 | '.11 Dissemination of findings | 22 |
| 8.0 | Ethical Considerations2 | 22 |
| 8.1 | Ethical committee approvals2 | 22 |
| 8 | 3.2 Risks & Benefits for Subjects | 23 |
| 8 | 3.3 Unexpected/Adverse Events | 23 |
| 8 | 3.4 Prevention of SARS-CoV-2 Infection in Investigation Personnel | 24 |
| 9.0 | Timeline2 | 25 |
| 10.0 | 0 Budget2 | 26 |
| 11.0 | O References | 27 |

| 12.0 Appendices |
|---|
| Appendix I: Participant Information Sheet - English |
| Appendix II: Participant Information Sheet - Bemba |
| Appendix III: Participant Information Sheet – Chewa/Nyanja |
| Appendix IV: SARS-CoV-2 ANC Surveillance Questionnaire |
| Appendix V: Other, e.g. permission letters |
| Appendix VI: C.Vs |

# Acronyms

| Acronym | Explanation |
|------------|-----------------------------------------------------------|
| ANC | Antenatal Care |
| CIDRZ | Centre for Infectious Disease Research in Zambia |
| CDC | U.S. Centers for Disease Control and Prevention |
| CHWs | Community Health Workers |
| COVID-19 | Coronavirus Disease |
| DHO | District Health Office |
| DBS | Dry Blood Spot |
| HIV | Human Immunodeficiency Virus |
| IRB | Institutional Review Board |
| MNCH | Maternal, Newborn and Child Health |
| МОН | Ministry of Health |
| MTA | Materials Transfer Agreement |
| NAAT | Nucleic Acid Amplification Test |
| NHRA | National Health Research Authority |
| ODK | Open Data Kit |
| PEPFAR | U.S. Presidential Emergency Plan for AIDS Relief |
| РНО | Provincial Health Office |
| PMTCT_STAT | Prevention of Mother to Child Transmission of HIV |
| PPE | Personal Protective Equipment |
| QA/QC | Quality Assurance/ Quality Control |
| SARS-CoV-2 | Severe Acute Respiratory Syndrome-Related Coronavirus-2 |
| SOPs | Standard Operating Procedures |
| UNZA BREC | University of Zambia Biomedical Research Ethics Committee |
| VTM | Viral Transport Media |
| ZNPHI | Zambia National Public Health Institute |

#### 1.0 Introduction

#### 1.1 General information on research topic

The novel coronavirus SARS-CoV-2, the cause of COVID-19, was first detected in Wuhan city, China in December 2019 and the first cases were confirmed in Zambia in March 2020. Current data suggest that as many as 50% of cases are asymptomatic [1]. Initial surveillance has focused primarily on patients with symptoms or severe disease, and, as such, the full spectrum of the disease, including the extent and fraction of mild or asymptomatic infections that do not require medical attention are not clear. Estimates of the case fatality ratio, and other epidemiological parameters, will likely be lower than current estimates once the full spectrum of disease is able to be included in the denominator. With any novel virus, such as SARS-CoV-2, initial population seroprevalence is assumed to be negligible. Thus, antibody seropositivity in a population can allow inferences to be made about the extent of infection, the cumulative incidence of infection in the population, and trends in infection over time.

This protocol proposes to investigate the extent of SARS-CoV-2 infection, as determined by seropositivity, among pregnant women attending 1<sup>st</sup> antenatal care (ANC) visits, as a surrogate for the prevalence in the general population. The utility of ANC-based surveillance has been established for malaria [2-5], and there is no evidence to date suggesting that pregnant women are at higher risk of contracting SARS-CoV-2 than non-pregnant adults, suggesting that ANC-based surveillance could provide useful information for monitoring the spread of SARS-CoV-2 over time [6]. This will be a non-randomized assessment of the potential to leverage pregnant women attending 1<sup>st</sup> ANC as a pragmatic sentinel population to monitor prevalence of SARS-CoV-2 and to detect changes in transmission in selected areas.

As the Zambian Ministry of Health (MOH) continues to focus on controlling and mitigating further spread of the SARS-CoV-2 through active surveillance for case detection, contact tracing, physical distancing and isolation while strengthening case-based management, it is important to build a national SARS-CoV-2 surveillance system that is crucial for containing transmission of the virus and preparing for future waves of the infection.

#### 1.2 Overview of research and research gaps

This surveillance platform may be able to provide key information on the spread of the SARS-CoV-2 virus through the general population. By using serologic testing to understand trends in the proportion of pregnant women over time who were exposed to SARS-CoV-2, we will be able to understand not only the ultimate proportion of pregnant women who were ever infected, but also be able to track and potentially detect outbreaks (e.g. in areas with increasing positivity rates), unlike data that would be available from a single cross-sectional survey, which could give the overall prevalence at a single point in time. In most places to date, testing has focused on symptomatic people, their contacts or others considered at high risk for infection, but there is limited understanding of the true proportion of asymptomatic cases.

There are gaps in information about the prevalence and clinical characteristics of SARS-CoV-2 in Zambia. We propose to conduct SARS-CoV-2 sentinel surveillance among first-time ANC attendees in selected Maternal, Newborn and Child Health (MNCH) departments in four districts (Lusaka, Chongwe, Chadiza and Chipata) of Lusaka and Eastern provinces to assess SARS-CoV-2 seroprevalence. Pregnant women will serve as a proxy for the healthy adult population of these districts, much as they have in sentinel surveillance for HIV and malaria. Because we will use serologic testing from blood and not nasal swabs, this collection will not substantially alter the risk for either the health worker nor the woman and will not deplete the supplies of SARS-CoV-2 Polymerase chain reaction (PCR) reagents used for diagnosis.

# 1.3 Overall purpose of the research

V4.1, 13 June 2021

The purpose of this project is to provide information on the seroprevalence of SARS-CoV-2 antibodies in the community with pregnant women as the sentinel population. CIDRZ will work with facility in-charges in the selected sentinel sites to provide sensitization and SARS-CoV-2 antibody testing to pregnant women presenting for their first ANC visit.

#### 2.0 Statement of the Problem

Zambia is experiencing a SARS-CoV-2 epidemic. From March 18, 2020 to February 19, 2021, at total of 73,203 confirmed cases have been reported in Zambia. However, the true number is likely much larger, because surveillance systems for SARS-CoV-2 in Zambia are incomplete [7]. ANC surveillance of SARS-CoV-2 antibodies could provide needed insights into transmission trends in the general population. This surveillance will provide a means to systematically detect SARS-CoV-2 antibodies in pregnant women and notify relevant authorities about the prevalence.

# 3.0 Rationale/ Justification

Since 2020, the coronavirus disease has become a major public health concern and sustainable and efficient surveillance platforms are urgently needed; assessing women attending 1<sup>st</sup> ANC should provide insights into transmission trends in the general population. This activity will determine what proportion of pregnant women demonstrate evidence of SARS-CoV-2 infection over time. The findings of this research may be used to change the way health system monitors the epidemic and ensures health services are made available with minimal disruptions.

#### 4.0 Literature Review

ANC surveillance has not been routinely utilized for SARS-CoV-2 in any country. A cross-sectional study from Cape Town, South Africa found a seroprevalence of 38% among residual serum from antenatal clinic attendees in July and August 2020 [8]. Six African countries including Zambia (i.e., Kenya, Malawi, Mozambique, Nigeria, Uganda, and Zambia) are piloting ANC surveillance based on experience for surveillance of other infectious diseases (HIV, syphilis, malaria) [9,10]. ANC surveillance has been a key strategy for HIV for many years, because women attending ANC clinics represent an accessible healthy population [11-13].

Prevalence estimates of SARS-CoV-2 infections have varied widely throughout Africa. This is likely a result of varying time, study population, and study design [14-20]. Nevertheless, SARS-CoV-2 infections are under-reported because of the large asymptomatic proportion of

infections, testing limitations, and surveillance gaps [21,22]. Africa is no exception, where several prevalence surveys (including in Zambia) have shown under-ascertainment of SARS-CoV-2 infections [7,23]. For instance, during a population-based study in six districts in Zambia in July 2020, the ratio of reported cases to estimated infections ranged from 1:1012 (Livingstone District) to 1:21 (Lusaka District) [7]; overall, only 1 case was reported for every 92 infections. In Cape Town, 5% of residual serum specimens from persons living with HIV and women attending ANC clinics testing positive for SARS-CoV-2 antibodies had positive PCR test results in the public health surveillance system [24]. Other studies from other African countries have revealed substantial under-ascertainment of SARS-CoV-2 infections [18,25-27]. Strategies for improvement in surveillance have been called for by the Africa CDC and others [28,29].

# 5.0 Research questions

This study will assess the seroprevalence of SARS-CoV-2 in pregnant women aged 15-49 years who present to the health facility for their first antenatal care visit. This surveillance will answer the following research question: "What is the seroprevalence of antibodies to SARS-CoV-2 among pregnant women attending first ANC visit in Zambia?"

#### 6.0 Research Aims and Objectives

#### 6.1 Research Aim

The primary aim of this activity is to determine SARS-CoV-2 seroprevalence from women attending antenatal clinics for their first ANC visit as an easy-access population for routine monitoring.

#### **6.2** Primary Objectives

- 6.2.1 To estimate on a monthly basis the seroprevalence of SARS-CoV-2 among pregnant women aged 15-49 years attending their first ANC visit at selected health facilities in Chadiza, Chipata, Chongwe, and Lusaka districts of Eastern and Lusaka Provinces.
- 6.2.2 To monitor trends in SARS-CoV-2 seroprevalence in the selected districts.

#### **6.3** Secondary Objectives

- 6.3.1 To determine the feasibility and acceptability of SARS-CoV-2 antibody tests among pregnant women
- 6.3.2 To estimate the prevalence of HIV-COVID 19 co-infection among pregnant women aged 15-49 years
- 6.3.3 To determine sociodemographic factors associated with SARS-CoV-2 seropositivity among pregnant women
- 6.3.4 To compare trends in seroprevalence among pregnant women with routine surveillance data to determine if ANC sentinel surveillance is a viable surveillance strategy for SARS-CoV-2

# 7.0 Methodology

#### 7.1 Study Design

This will be a passive surveillance of pregnant women attending their first antenatal care visit at the selected study sites in the four selected districts. Pregnant women attending 1st ANC will be used as a pragmatic sentinel population to monitor the seroprevalence of SARS-CoV-2 over time. Women will be informed of this activity during group health education sessions and will be consented during individual HIV testing and counselling. To minimize discomfort to the participant, spots of blood will be collected from all women consenting to participate (up to 20 women per study site per month) on filter paper for a SARS-CoV-2 serologic test using a finger prick or a venous blood draw, depending on the method being used to obtain blood for routine HIV and syphilis testing during first ANC visits. In addition, women will be asked to respond to a short questionnaire. The woman's name will not be included on the sample or on the form; rather, a unique study ID will be used to link the questionnaire to the sample. Seroprevalence data will be aggregated at the district level on a monthly basis.

#### 7.2 Study Site and Population

#### 7.2.1 Study Sites

Study sites will be selected in each of four purposively selected districts using a probabilityproportional-to-size selection of 10 eligible facilities within each district. Eligible facilities will have averaged at least 19 first ANC visits per month over the course of the previous year. Surveillance activities will be implemented in two urban and rural districts as follows:

Table 1: Study sites and sampling interval for SARS-CoV-2 seroprevalence surveillance in ANC clinics in Chadiza, Chipata, Chongwe, and Lusaka Districts - Zambia

| District | | Facility | Average<br>monthly ANC<br>attendance<br>(2020)* | Sampling<br>interval |
|---|---|---|---|---|
| Chadiza | 1 | Chanida Rural Health Centre | 19 | 1 |
| | 2 | Nsadzu Rural Health Centre | 21 | 1 |
| | 3 | Madzaela Health Post | 21 | 1 |
| | 4 | Bwanunkha Rural Health Centre | 23 | 1 |
| | 5 | Chanjowe Health Post | 24 | 1 |
| | 6 | John Rural Health Centre | 24 | 1 |
| | 7 | Mkumbuzi Rural Health Centre | 28 | 1 |
| | 8 | Zemba Rural Health Centre | 36 | 1 |
| | 9 | Chadiza Rural Health Centre | 44 | 2 |
| | 10 | Miti Rural Health Centre | 46 | 2 |
| Chipata | 1 | Champhande Rural Health Centre | 21 | 1 |
| | 2 | Chikando Rural Health Centre | 23 | 1 |
| | 3 | Lunkwakwa Urban Health Centre | 25 | 1 |
| | 4 | Mwami Hospital Affiliated Health<br>Centre | 28 | 1 |
| | 5 | Chipata Hospital Affiliated Health<br>Centre | 34 | 1 |
| | 6 | Jerusalem Rural Health Centre | 35 | 1 |
| | 7 | Walela Health Post | 56 | 2 |
| | 8 | Mchini Health Post | 69 | 3 |
| | 9 | Namseche Rural Health Centre | 92 | 4 |
| | 10 | Kapata Urban Health Centre | 162 | 8 |
| Chongwe | 1 | Nchute Health Post | 19 | 1 |
| | 2 | Chikumbi Health Post | 22 | 1 |
| | 3 | Kasisi Rural Health Centre | 23 | 1 |
| | 4 | Palabana Rural Health Centre | 24 | 1 |
| | 5 | Kanakantapa Rural Health Centre | 27 | 1 |
| | 6 | Water Falls Rural Health Centre | 28 | 1 |
| | 7 | Katoba Rural Health Centre | 32 | 1 |
| | 8 | Chainda Rural Health Centre | 35 | 1 |
| | 9 | Ngwerere Main Rural Health Centre | 109 | 5 |
| | 10 | Chongwe Referral Rural Health Centre | 137 | 6 |
| Lusaka | 1 | Coptic Hospital | 21 | 1 |
| | 2 | Kuku Health Post | 98 | 4 |
| | 3 | Chainda Urban Health Centre | 99 | 4 |
| | 4 | Matero Main Urban Health Centre | 228 | 11 |

| | 5 | Chaisa Urban Health Centre | 231 | 11 |
|---|---|---|---|---|
| | 6 | Kanyama West Health Post | 246 | 12 |
| | 7 | George Urban Health Centre | 371 | 18 |
| | 8 | Matero First Level Hospital | 407 | 20 |
| | 9 | Kanyama First Level Hospital | 572 | 28 |
| | 10 | University Teaching Hospital - Adult | 606 | 30 |
| * Based upon PMTCT_STAT indicator from PEPFAR MER | | | | |

#### **7.2.2** Study Population

A sample of 20 pregnant women attending their first ANC visit at the selected study sites will be enrolled into the study until the monthly sample size is reached.

# 7.3 Selection of Participants, Sampling and Sample Size

#### 7.3.1 Selection of Participants

Women presenting to the selected study sites for their first ANC visit at selected health facilities in the four districts will be eligible to participate in the study. A facility-specific interval for systematic sampling will be defined based on each facility's monthly mean number of women attending their first ANC visit based on the historic monthly ANC attendance during fiscal year 2020. until the monthly sample size is met at a given facility. Data will be collected over a 12-15 months period of implementation to ensure that the number of required samples are met in all implementing sites.

#### 7.3.1.1 Inclusion criteria

All women presenting to the selected study sites will be considered for inclusion into the study if they are:

- Confirmed pregnant and are registered for their first ANC visit
- Aged 15 to 49 years
- Able to provide consent to participate and have blood sample collected for the SARS-CoV-2 antibody test

#### 7.3.1.2 Exclusion criteria

- Not first ANC visit for the pregnant woman
- Women less than 15 years or above 49 years old
- Women not able to provide consent for study participation

#### 7.3.2 Sample Size

All pregnant women who meet the eligibility criteria presenting at the study sites will be approached for participation into the study. Monthly ANC attendance varies by district, as shown in Table 2. Study districts will be expected to recruit 200 pregnant women per month. The estimated seroprevalence is expected to vary by study site, as prevalence has been demonstrated to be different between urban and rural locations in Zambia [7]. A sample size of 200 women per district per month will be sufficient to detect a range of estimated proportions of SARS-CoV-2 seroprevalence (Figure 1). The confidence interval (CI) reflects the bounds of the true seroprevalence of COVID-19 among pregnant women attending ANC (and not the overall pregnant women population or general population). Where prevalence is expected to be low (i.e. rural districts), a sample size of 200 women produces a 95% CI half-width of 2.4% for 3% seroprevalence (lowest estimate). Where prevalence is expected to be higher (i.e. urban districts), a sample size of 200 women produces a 95% CI half-width of 7.0% for 50% seroprevalence. Women will be recruited evenly throughout the month from study sites selected for each district. If the monthly recruitment target is met, study sites will be expected to pause sample collection and reconvene at the start of the next month.

| Table 2: Average monthly number of | |
|--------------------------------------|-----------------|
| first ANC attendees using PMTCT_STAT | |
| denominator | |
| District | Average monthly |
| | ANC attendance |
| Chadiza | 424 |
| Chipata | 759 |
| Chongwe 653 | |
| Lusaka | 6,378 |



#### 7.4 Implementation of Procedures

#### 7.4.1 Implementation of pre-survey activities

# 7.4.1.1 Engage and mobilize stakeholders

At the beginning of the study, we will systematically identify and engage stakeholders (Provincial and District Health Offices (PHO/DHOs) and other implementing partners) to help build involvement and allow them to participate in the planning of activities for implementation and ensure that their expectations are met.

#### 7.4.1.2 Community engagement and sensitization

Information about the study will be cascaded to various levels of the community through sensitizations meetings with community leaders such as headmen, teachers and political leaders. Health care providers at all the sentinel sites will be part of the sensitization meetings with the community. Additionally, information about the study will be incorporated in routine health talks which are given to pregnant women as they come to register for ANC.

#### 7.4.1.3 Train DHO staff from sentinel sites

Health facility in-charges and healthcare workers from the MNCH departments and laboratory hubs will be oriented in the approved study protocol by MOH/CIDRZ research teams and supported throughout the study time. They will also be trained in phlebotomy/specimen collection, labeling and storage, biohazard waste disposal, transfer of specimens, and quality assurance and control. Study staff will also be trained in data collection, documentation, storage and safety, reporting and monitoring. All staff participating in implementation of study activities will be required to obtain good clinical practice and human research protection training. Laboratory staff will be reoriented on running of assays to be used in the study. Additionally, on-site orientation will be conducted to enhance hands-on experience of study procedures. Lay healthcare providers and Peer Educators who have been providing support at the study sites will be selected and trained to provide support for study specific tasks such as participant identification and provision of health education. All staff will be provided with SOPs which will provide them step-by-step instructions on how to perform study procedures.

#### 7.4.1.4 Develop data collection and management tools

The following standard operating procedures will be developed to provide written step-by-step instructions to help study staff to perform routine tasks at the study sites: screening and eligibility, informed consent, study enrolment, sample collection, handling and testing, data collection and management (questionnaire completion, data entry, security, QA/QC), roles and responsibilities SOP, etc).

In addition, a basic questionnaire will be used to collect information from consented ANC attendees. This questionnaire contains information about symptoms of COVID-19, possible exposures to SARS-CoV-2, and risk mitigation behaviors. Additionally, the questionnaire will collect information on sociodemographic characteristics and routine ANC lab results (HIV, syphilis, Hepatitis B, and malaria).

#### 7.4.1.5 Procure study supplies

Study sites will be supplied with all required commodities (i.e., assays, lancets, handwarmers, microtainers, dry blood spot (DBS) cards, protective clothing, polyester fiber-tipped applicator, paper towel, waste segregation polythene bag, depressors, cool box, ice packs, bleach, hand sanitizer, scissors, cryovial with virus transport media (VTM), a fine tipped permanent marker, barcodes, bar code scanner, specimen collection and transportation log forms, etc.) to enable them to collect DBS samples for the SARS-CoV-2 serologic tests. The study will outsource tablets for data entry purposes. Laboratories will be equipped with all necessary materials to process and run DBS samples.

#### 7.4.2 Implementation of survey activities

#### 7.4.2.1 Recruitment of study participants

All study processes will be undertaken as part of routine ANC so as not to disrupt patient flow. Women will be informed of this activity during group health education at the beginning of the first ANC visit. Health education on SARS-CoV-2 will cover symptoms of active infection, testing, and prevention methods, but will emphasize that this study looks for antibodies to SARS-CoV-2 in the blood which are NOT an indicator of current infection.

Women experiencing symptoms of COVID-19 will be managed according to national guidelines (such women will not be recruited in the study because they will not proceed with routine ANC given their acute complaints). Women will be informed that the quality of their antenatal care will not be impacted by their decision whether or not to participate in the study. If they do participate, they will not receive their test results as this study aims to measure population level seroprevalence and does not impact individual clinical care. Women will be approached for consent during individual counseling and testing sessions and blood will be collected on filter paper for a SARS-CoV-2 serologic test using blood from the same finger prick as that for HIV and syphilis testing. While waiting for HIV test results, consenting women will be asked to respond to a short questionnaire. Study participants will then continue with the remainder of the ANC visit as usual.

Sites should have regular access to serological and other routine tests required for care of pregnant women. As a test of past infection, serology results will not be communicated to the facility or participants because they do not affect clinical care (i.e. vaccine eligibility). Any woman that has symptoms of COVID-19 will be referred to relevant testing facility and will follow the national SARS-CoV-2 testing and treatment guidelines. Because they will receive evaluation for their acute complaints per national guidelines, they will not undergo routine ANC services, and, thus, will not be eligible for participation in this study.

#### 7.4.2.2 Sample collection, labelling, storage and courier

All staff (i.e., study and health facility staff) involved in the collection and transportation of specimen will be trained in safe handling practices and spill decontamination procedures. After obtaining consent from the participant and completing the study questionnaire and while maintaining rapport with the participant, the research nurse or phlebotomy staff will collect blood samples onto a dry-blood spot (DBS) card using finger stick procedures by trained staff. DBS samples collected on filter paper using a standard operating procedure will be used for SARS-CoV-2 antibody detection. Specimen and questionnaires will be labeled at time of collection with an identification sticker that has a pre-printed unique study ID and laboratory specimen ID, and current date. A paper log will be completed by study staff that contains the date, study staff ID, study ID, and a lab label to create a paper

trail in case of mislabeling. This paper log will be stored at the health facility and collected by the study team on a monthly basis. DBS cards will be placed in a bag prior to transportation to district hub laboratories for storage and testing using the existing viral load sample courier system supported by PEPFAR.

DBS cards will be tested for anti-SARS-CoV-2 antibodies using a serologic assay. The specific assay has not been determined yet, as potential cross-reactivity is an emerging issue in Africa [30,31]. Ongoing studies at CDC in Atlanta will inform assay selection. Analyses will be done at a hub or central laboratory. Samples will be kept until the study procedures outlined in the protocol are completed or for up to three years, at which time any remaining samples will be destroyed. The samples will not be used for another purpose than what is stated in the protocol.

Sample analysis will be batched as appropriate; total antibodies or IgG antibodies to SARS-CoV-2 will be assessed using laboratory-based serological assays such as enzyme linked immunosorbent assay (ELISA), immunofluorescence (IFA), chemiluminescent assays (CLIA), multiplexed bead-based assays (the specific assay to be utilized in the study in pending guidance from CDC in Atlanta). All testing will be conducted under appropriate and recommended biosafety conditions per CDC guidance.

# 7.5 Quality control and Assurance activities (supervisory, data and logistics monitoring)

Project supervisors will review the data collection forms and aggregate results on a monthly basis to assess for completeness, accuracy, and consistency. Periodic site visits will be conducted by the research team to assess for adherence to protocol procedures. Deviation from study protocols will be documented in an incident report and reported to the IRB within three working days. Additionally, up to 20% of samples may be run in duplicate at a central laboratory in Lusaka for the purposes of quality assurance.

# 7.6 Study staff roles and responsibilities

CIDRZ will support the Ministry of Health/Zambia National Public Health Institute to undertake this surveillance by providing technical assistance, training and mentoring of staff based in the health facilities and DHOs, project oversight, and supplies procurement. The project may be supplemented by PEPFAR funded activities as well as with additional technical support from CDC Zambia. The roles and responsibilities of CIDRZ supported are as outlined:

#### 7.6.1 Technical Lead

The technical lead will be responsible for technical oversight throughout the study period. Before implementation, the technical lead will lead protocol development and submission for ethical approval. The technical lead will participate in developing SOPs and training study staff as well as monitoring data reporting and quality control activities. Upon completion of the study, the technical lead will coordinate preparation and dissemination of the final report.

#### 7.6.2 Study Coordinator

The study coordinator will support study implementation by ensuring that all study activities are being implemented as laid out in the approved protocol. He/she will prepare the ethics application and ensure that study staff are working in compliance with, and be responsible for, tracking the project milestones. The study coordinator will manage the study budget, provide support for recruiting and training of staff. Additionally, he/she will be the point of contact between the principal investigator and staff at study sites.

#### 7.6.3 Research Nurse

One research nurse will be employed for each of the study sites. Their role will be to ensure site compliance with the approved protocol by reviewing regulatory requirements. They will be responsible for communicating information about the study to potential participants and ensuring that staff involved with study implementation have the correct credentials and study related training. The research nurse will draw a blood sample onto filter paper via finger prick for SARS CoV-2 antibody testing and will adhere to sample storage and

transportation procedures. They will also ensure that correct source documents are used and that data is accurately captured in the questionnaires. They will act as the point of contact between the study coordinator and site staff.

#### 7.6.4 Community Health Workers

Community health workers advocate for underserved communities to receive services and will be engaged from the already existing cadres known at the facility to supplement efforts of MOH HCWs and research nurses. For this study, they will conduct health education to pregnant women attending ANC visits. They will also be trained on how to collect information from the ANC attendees and administer the questionnaire.

#### 7.6.5 Data Coordinator

The data coordinator will provide support for data management. He/she will ensure that ANC COVID folder on the central server is updated routinely and resolve any problems with the database. He will conduct quality improvement activities and liaise with the study coordinator about any identified quality problems with the data.

#### 7.6.6 Program Assistant

The program assistant will provide administrative support for the study. He/she will submit request for supply purchases, make regular follow ups about delivery timelines and keep stock of supplies. In addition, he/she will submit cash requests for various activities and ensure that receipts are submitted to the Finance office as per stipulated guidelines. The program assistant will identify venues for trainings and communicate with the vendor about scheduled trainings.

# 7.7 Data collection and management

The study questionnaire and database will be designed using Open Data Kit (ODK)—a free, open-source suite of tools that will allow collection of data using android mobile devices without Internet connectivity. CHWs will be trained to administer the electronic questionnaire that will be uploaded onto password protected android devices (see appendix IV) which will be piloted to ensure that data is correctly captured and stored when data

collection begins. Individual respondents will be assigned a unique identifier to assist with data confidentiality. Respondents' names and other personally identifying information will not be recorded in the questionnaire. Data will be uploaded to a server after each day of ANC data collection. Data collection devices (tablets, storage card) will be handled only by facility or study staff and kept in a locked office, in a lockable cabinet. Data will be exported to MS Excel for cleaning once every week. Any missing variables will be communicated to the research nurse for follow up and action with the CHW.

#### 7.8 Data analysis

Data will be analyzed on a monthly basis using a statistical program. Basic descriptive statistics, by district, including prevalence point estimates, confidence intervals, and relative standard errors will be tabulated. Variance and confidence intervals will be adjusted for health facility clustering. Prevalence estimates will be disaggregated by sociodemographic variables, routine ANC lab results, and risk factors.

#### 7.9 Data Ownership

All data collected through this protocol are the property of the Zambian Ministry of Health. All reviews and decisions regarding data sharing, for example at the request of a journal at the time of publication, will be made by the MoH as the owners of the primary data according to NHRA policies and procedures.

#### 7.10 Sponsor monitoring

CDC is the primary sponsor for the activities described herein. As the sponsor, the CDC may conduct monitoring or auditing of activities to ensure the integrity of the data collected and to ensure the rights and protection of individuals. Monitoring and auditing activities may be conducted by:

- 7.10.1 CDC staff ("internal")
- 7.10.2 Authorized representatives of CDC (e.g., a contracted party considered to be "external")
- 7.10.3 Both internal and external parties.

Monitoring or auditing may be performed by means of on-site visits to government facilities or through other communications such as telephone calls or written correspondence. The visits will be scheduled at mutually agreeable times, and the frequency of visits will be at the discretion of CDC. During the visit, any related materials may be reviewed and the CoAg along with the relevant staff should be available for discussion of findings. To ensure compliance with national and international regulatory guidelines, the activities outlined in this proposal may be subject to inspection or review by authorized Zambian or international regulatory authorities, including the UNZA BREC, NHRA, and US IRBs.

## **7.11** Dissemination of findings

Monthly summary data from the ANC visits at all participating facilities will be monitored to ensure that data are being collected correctly, however, no formal interim analyses will be conducted. Results will be presented by CIDRZ through tables and disseminated through reports to the Ministry of Health, ZNPHI, CDC, and other stakeholders. Results will also be disseminated through conference presentations and through publications in peer reviewed journals.

#### 8.0 Ethical Considerations

#### 8.1 Ethical committee approvals

The study protocol will be reviewed by the local IRB (UNZA BREC) and CDC before data collection starts for appropriate input and approvals. An information sheet with details about the study will be offered to eligible participants in their preferred language (i.e., (Chewa/Nyanja, Bemba) while study staff provide detailed explanation about the study procedures Participants will be told the general purpose, the possible risks, and benefits in the local language (Nyanja/Chewa or Bemba). Individual written consent will be obtained before sample collection and administration of the questionnaire. Pregnant and recently pregnant women are considered emancipated minors for the purpose of providing their own informed consent. Women will be offered a copy of the consent form if they wish to take it. Participation is voluntary and refusal will not affect a participant's health care. Additionally, participants may refuse to answer specific questions during the questionnaire.

# 8.2 Risks & Benefits for Subjects

This investigation poses minimal risk to participants, involving the collection of a small amount of blood. Every attempt will be made to utilize the finger prick being made for routine HIV and syphilis testing during the first ANC visit. During the blood collection, women may experience temporary discomfort, and there is a very small risk of infection. The area will be cleaned thoroughly prior to drawing blood to prevent infection. There are no economic risks associated with this study. Pregnant women will not be asked to make any additional visits to the health facility specifically for the purposes of the study. However, the participants may spend additional time (estimated 10 minutes) at the facility during the first ANC visit to complete the questionnaire. The primary benefit of the study is indirect in that data collected will help improve and guide efforts to understand the extent of SARS-CoV-2 infection, which might help contribute to efforts to prevent further transmission of the virus in Zambia. There is no specific direct benefit to participants.

Of note, this activity will NOT contribute to clinical care of the participants in real-time. Among other reasons, this is because serologic conversion in general does not occur until after acute illness; because serologic tests are not diagnostic for current SARS-CoV-2 infection, they are inappropriate for clinical decision making; and because lab analysis would take place remotely and results would not be available until at best days or weeks after the clinic visit. Further, as we will not record any identifiers on the filter paper samples, it will not be possible to link the results of SARS-CoV-2 serologic testing back to the woman from whom the sample was taken.

#### 8.3 Unexpected/Adverse Events

This study does not entail substantial risk to any participants. However, any major deviations from the protocol will be treated as an unanticipated problem/event and will be reported to all IRBs of record within the timeframe specified by the IRB. This also includes any problem or event that: 1) poses harm or risk of harm to subjects or others; 2) is unanticipated (not described in research plan or consent form); and 3) related to the study procedures.

# 8.4 Prevention of SARS-CoV-2 Infection in Investigation Personnel

All personnel involved in the investigation will be trained in infection prevention and control procedures for SARS-CoV-2 as detailed by the Zambian Ministry of Health, including proper correct use of masks, physical distancing, limiting time in enclosed and/or crowded spaces, and hand hygiene. Personnel who develop symptoms will be isolated, tested, and referred appropriately. They will be allowed to resume involvement after resolution of symptoms and completion of recommended days in isolation.

V4.1, 13 June 2021

# 9.0 Timeline

| A saturation | Danie a sible Danie | Duration in Months | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Activities | Responsible Person | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 |
| Adaptation of protocol to UNZA BREC | PI/Technical Lead | Х | | | | | | | | | | | | | | |
| Submission and approval | PI/ Technical Lead | | Х | | | | | | | | | | | | | |
| Training for all DHO staff and facility in charges from sentinel sites | Technical Lead/ Study<br>Coordinator | | | Х | | | | | | | | | | | | |
| On site orientation for all MCH staff in the sentinel sites | Study Coordinator/<br>Study Nurses | | | Х | | | | | | | | | | | | |
| Enrolment of participants | Facility Staff/<br>Study Nurses | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Supervisory visits to sentinel sites | All | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Monitoring availability of all logistics and surveillance activities | Study Coordinator/<br>Study Nurses/<br>Program Admin | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Monthly data reporting and monitoring | Study Nurses | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Quality control and assurance activities | Technical Lead/ Study<br>Coordinator | | | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х |
| Data analysis and preparation of the final report | Technical Lead/ SI team | | | | | | | | | | | | | | Х | Х |
| Presentation of final report by CIDRZ to MoH<br>Senior staff, ZNPHI and CDC | PI/ Technical Lead | | | | | | | | | | | | | | | Х |
| Presentation of the results by MoH/ZPHI to various stakeholders | MoH/AII | | | | | | | | | | | | | | | Х |
| Submission of the copy of report to Scientific and Ethical Committee | Technical Lead | | | | | | | | | | | | | | | Х |
| Dissemination of findings (Journal publication, abstract and poster) | Technical Lead | | | | | | | | | | | | | | | Х |
| Posting findings on Government and CIDRZ websites | Technical Lead | | | | | | | | | | | | | | | Х |

# 10.0 Budget

We are requesting a total of US\$300,992.02 which will be allocated to personnel, travel, supplies and other costs. The budget has been broken down as follows:

| | Category | Cost (US\$) | % |
|-----------|-------------------------------------------|-------------|-------|
| Personnel | | 60,897.93 | 20.23 |
| Equipment | | - | - |
| Supplies | | 125,366.00 | 41.66 |
| Travel | | 42,120.00 | 13.99 |
| Other | | | 24.12 |
| | Trainings | 26,508.07 | |
| | Stakeholder meetings | 1,500.00 | |
| | Communication | 3,600.00 | |
| | Administrative costs | 9,000.00 | |
| | Stipends for ANC TS and transport refunds | 35,000.00 | |
| CIDRZ IDC | | - | |
| Total | | 300,992.01 | 100 |

#### 11.0 References

- 1. Oran DP, Topol EJ. Prevalence of Asymptomatic SARS-CoV-2 Infection: A Narrative Review. Ann Intern Med. 2020 Sep 1;173(5):362-367. doi: 10.7326/M20-3012. Epub 2020 Jun 3. PMID: 32491919; PMCID: PMC7281624.
- 2. van Eijk, A.M., et al., Prevalence of malaria infection in pregnant women compared with children for tracking malaria transmission in sub-Saharan Africa: a systematic review and meta-analysis. The Lancet Global Health, 2015. 3(10): p. e617-e628
- 3. Hellewell, J., et al., Using ante-natal clinic prevalence data to monitor temporal changes in malaria incidence in a humanitarian setting in the Democratic Republic of Congo. Malar J, 2018. 17(1): p. 312.
- 4. Kitojo, C., et al., Estimating malaria burden among pregnant women using data from antenatal care centres collected between 2014 and 2017 and implications for elimination strategies in Tanzania: a population-based study Lancet Global Health, 2019.
- 5. Willilo, R.A., et al., Pregnant women and infants as sentinel populations to monitor prevalence of malaria: results of pilot study in Lake Zone of Tanzania. Malar J, 2016. 15(1): p. 392.
- 6. National Center for Immunization and Respiratory Diseases, Division of Viral Diseases. COVID-19: Pregnancy, Breastfeeding, and Caring for Newborns. Centers for Disease Control and Prevention, 28 Dec. 2020. <a href="https://www.cdc.gov/coronavirus/2019-ncov/need-extra-precautions/pregnancy-breastfeeding.html">https://www.cdc.gov/coronavirus/2019-ncov/need-extra-precautions/pregnancy-breastfeeding.html</a>
- 7. Mulenga LB, H.J., Fwoloshi S, et al., *Prevalence of Severe Acute Respiratory Syndrome*Coronavirus 2 (SARS-CoV-2) Infection in Six Districts in Zambia—July 2020: a cross-sectional multi-stage cluster-sampled household survey. Lancet Glob Health, 2021.

https://www.thelancet.com/journals/langlo/article/PIIS2214-109X(21)00053-X/fulltext

- 8. National Institute for Communicable Diseases. SARS-CoV-2 seroprevalence in the Cape Town Metropolitan Subdistricts after the peak of infections. COVID-19 Spec Public Heal Surveill Bull. 2020;18(Supplementary issue 5):1–9. <a href="https://www.nicd.ac.za/wp-content/uploads/2020/09/COVID-19-Special-Public-Health-Surveillance-Bulletin Issue-5.pdf">https://www.nicd.ac.za/wp-content/uploads/2020/09/COVID-19-Special-Public-Health-Surveillance-Bulletin Issue-5.pdf</a>
- 9. Kamocha S, Mulenga C, Mwakazanga D, Monze M, Nyoni I, Soud F, Shields M, Marx M. Declining HIV prevalence in Zambia: sentinel surveillance programmatic insight and the

need for HIV incidence data. Sex Transm Infect July 2013 Vol 89 (Suppl 1):A1–A428. https://sti.bmj.com/content/sextrans/89/Suppl 1/A212.2.full.pdf

- 10. Kangale C, Musunse M, Phiri-Chibawe C, Hamainza B, Psychas, P, Heilmann L, Miller JM, Gutman JR. Assessing malaria prevalence and intervention coverage from routine antenatal care visits in Chadiza District, Eastern Province, Zambia. ASTMH 2020. LB-5073
- 11. Guidelines for conducting HIV sentinel serosurveys among pregnant women and other groups/UNAIDS/WHO Working Group on Global HIV/AIDS and STI Surveillance. 2003; Geneva, Switzerland: Joint United Nations Programme on HIV/AIDS (UNAIDS) and World Health Organization (WHO), 66.

https://www.who.int/hiv/pub/surveillance/en/ancguidelines.pdf?ua=1

- 12. Eaton JW, Rehle TM, Jooste S, Nkambule R, Kim AA, Mahy M, Hallett TB. Recent HIV prevalence trends among pregnant women and all women in sub-Saharan Africa: implications for HIV estimates. AIDS. 2014 Nov;28 Suppl 4(4):S507-14.
- 13. UNAIDS/WHO working group on global HIV/AIDS and STI surveillance. Conducting HIV surveillance based on routine programme data among pregnant women attending antenatal clinics. August 2015.

https://www.unaids.org/sites/default/files/media asset/SurveillanceRoutineProgrammeDat a en.pdf

- 14. Alemu BN, Addissie A, Mamo G, et al. Sero-prevalence of anti-SARS-CoV-2 Antibodies in Addis Ababa, Ethiopia. bioRxiv [Internet]. 2020;2020.10.13.337287. Available from: <a href="http://biorxiv.org/content/early/2020/10/13/2020.10.13.337287.abstract">http://biorxiv.org/content/early/2020/10/13/2020.10.13.337287.abstract</a>
- 15. Majiya H, Aliyu-Paiko M, Balogu VT, et al. Seroprevalence of COVID-19 in Niger State. medRxiv [Internet]. 2020;(June):2020.08.04.20168112. Available from:

https://www.medrxiv.org/content/10.1101/2020.08.04.20168112v1%0Ahttps://www.medrxiv.org/content/10.1101/2020.08.04.20168112v1.abstract

16. Shaw J, Meiring M, Cummins T, et al. Higher SARS-CoV-2 Seroprevalence in Workers with Lower Socioeconomic Status in Cape Town, South Africa. [Internet]. Research Square. 2020. Available from: <a href="https://assets.researchsquare.com/files/rs-136543/v1/5bc4a4d1-031c-476b-b2b7-7a23da2577d6.pdf">https://assets.researchsquare.com/files/rs-136543/v1/5bc4a4d1-031c-476b-b2b7-7a23da2577d6.pdf</a>

- 17. Chibwana M, Jere K, Kamng'ona R, et al. High SARS-CoV-2 seroprevalence in health care workers but relatively low numbers of deaths in urban Malawi. medRxiv [Internet]. 2020; Available from: <a href="https://www.medrxiv.org/content/10.1101/2020.07.30.20164970v3">https://www.medrxiv.org/content/10.1101/2020.07.30.20164970v3</a>
- 18. Uyoga S, Adetifa IMO, Karanja HK, et al. Seroprevalence of anti–SARS-CoV-2 IgG antibodies in Kenyan blood donors. Science (80- ). 2020;eabe1916.
- 19. Halatoko WA, KONU YR, Gbeasor-Komlanvi FA, et al. Prevalence of SARS-CoV-2 among high-risk populations in Lomé (Togo) in 2020. *medRxiv* 2020.
- 20. Olayanju O, Bamidele O, Edem F, et al. SARS-CoV-2 Seropositivity in Asymptomatic Frontline Health Workers in Ibadan, Nigeria. *Am J Trop Med Hyg* 2020.
- 21. Bajema, K.L., et al., *Estimated SARS-CoV-2 Seroprevalence in the US as of September 2020.* JAMA Intern Med, 2020.
- 22. Pullano, G., et al., *Underdetection of cases of COVID-19 in France threatens epidemic control.* Nature, 2021. **590**(7844): p. 134-139.
- 23. Ojal J, B.S., Were V, et al., Revealing the extent of the COVID-19 pandemic in Kenya based on serological and PCR-test data. 2020: medRxiv [Internet]. . p. 1-32.
- 24. National Institute for Communicable Diseases. SARS-CoV-2 seroprevalence in the Cape
  Town Metropolitan Subdistricts after the peak of infections. COVID-19 Spec Public Heal
  Surveill Bull. 2020;18(Supplementary issue 5):1–9. <a href="https://www.nicd.ac.za/wp-content/uploads/2020/09/COVID-19-Special-Public-Health-Surveillance-Bulletin Issue-5.pdf">https://www.nicd.ac.za/wp-content/uploads/2020/09/COVID-19-Special-Public-Health-Surveillance-Bulletin Issue-5.pdf</a>
- 25. High SARS-CoV-2 seroprevalence in health care workers but relatively low numbers of deaths in urban Malawi. *medRxiv*. 2020; (published Aug 5.) (preprint).

#### https://doi.org/10.1101/2020.07.30.20164970v3

- <u>26.</u> NCDC and NIMR Release Findings of COVID-19 Household Seroprevalence Surveys in Four States of Nigeria. [Press Release] 22 February 2021.
- https://reliefweb.int/report/nigeria/ncdc-and-nimr-release-findings-covid-19-household-seroprevalence-surveys-four-states
- 27. 1 million people already exposed to COVID-19 in Accra, scientists estimate. [Press Release] <a href="https://www.waccbip.org/1-million-people-already-exposed-to-covid-19-in-accrascientists-estimate/">https://www.waccbip.org/1-million-people-already-exposed-to-covid-19-in-accrascientists-estimate/</a>
- 28. Massinga Loembé M, Tshangela A, Salyer SJ, Varma JK, Ouma AEO, Nkengasong JN. COVID-19 in Africa: the spread and response. Nat Med. 2020 Jul;26(7):999-1003.

- 29. Usuf E, Roca A. Seroprevalence surveys in sub-Saharan Africa: what do they tell us? Lancet Glob Health. 2021 Mar 9:S2214-109X(21)00092-9.
- 30. Tso FY, Lidenge SJ, Peña PB, et al. High prevalence of pre-existing serological cross-reactivity against SARS-CoV-2 in sub-Sahara Africa. Int J Infect Dis [Internet]. 2020
  31. Yadouleton A, Sander AL, Moreira-Soto A, et al. Limited Specificity of Serologic Tests for

SARS-CoV-2 Antibody Detection, Benin. *Emerg Infect Dis* 2020;27(1).